CLINICAL TRIAL: NCT06514209
Title: Effect of Different Depths of Neuromuscular Blockade on Respiratory Mechanics in Patients With Moderate-severe Acute Respiratory Distress Syndrome
Acronym: ARDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Lihong Xu, Resident physician, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARDS-NMBAs study 2024-07-09
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: ARDS; Lung Protective Ventilation
Keywords: ARDS; lung protective ventilation; neuromuscular blockade; respiratory mechanics
MeSH Terms: interventions — cisatracurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderate-Severe ARDS patients (Experimental): The dose of cisatracurium was gradually adjusted to achieve different depth of muscle relaxation
  Interventions: Drug: cisatracurium

INTERVENTIONS:
Drug: cisatracurium — The initial bolus dose of cisatracurium injection is 0.05-0.1mg/kg, followed by a continuous infusion of 1ug/kg/min of cisatracurium, with data on vital signs, respiratory mechanics, TOF response, etc. recorded after a 15-minute wait. The maintenance infusion dose of cisatracurium is then gradually increased in a gradient of 0.5ug/kg/min, with data collection after a 15-minute wait after each increase. If the patient's spontaneous breathing completely disappears, the infusion dose of cisatracurium will no longer be increased, and the titration will end.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is characterized by acute diffuse alveolar injury caused by a variety of pulmonary and extrapulmonary factors, leading to refractory hypoxemia. It has high incidence and mortality rates. Neuromuscular blocking agents (NMBAs) play a crucial role as adjunctive therapy for ARDS, aiding in lung-protective ventilation by inhibiting excessive spontaneous breathing, improving patient-ventilator synchrony, and reducing barotrauma.

Determining the appropriate depth of muscle relaxation in moderate to severe ARDS patients receiving NMBAs remains a clinical challenge. Research has shown that partial neuromuscular blockade is feasible in certain ARDS patients. However, large randomized controlled trials (RCTs) and clinical practices often use higher doses of NMBAs to ensure complete cessation of spontaneous breathing. This indicates an ongoing debate regarding the optimal depth of neuromuscular blockade necessary for lung-protective ventilation in ARDS patients. It also raises the question of whether the optimal depth of neuromuscular blockade varies among patients with different severities of ARDS.

This study aims to investigate changes in respiratory mechanics and other physiological parameters in moderate to severe ARDS patients under different depths of neuromuscular blockade. The investigators will evaluate the impact of targeted neuromuscular blockade depth on lung protection in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe ARDS requiring the use of NMBAs, as assessed by clinicians (Berlin definition 2012: PaO2/FiO2 < 150 mmHg, PEEP ≥ 5).
2. Age: 18-85 years.
3. Signed informed consent.

Exclusion Criteria:

1. History of allergy to NMBAs.
2. Open chest or abdominal injuries.
3. Patients with pulmonary masses, lung transplantation, or lung resection.
4. Contraindications to esophageal catheter placement.
5. Pregnant patients.
6. Contraindications to TOF measurement (e.g., history of neuromuscular disease, presence of a cardiac pacemaker).
7. Severe dysfunction of other organs with an expected short-term mortality (within 7 days) or palliative care.
8. Previous inclusion in this study.

Ages: 18 Days to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
transpulmonary pressure (PL) | At baseline and 15 minutes after each adjustment of the cisatracurium dose.

SECONDARY OUTCOMES:
esophageal pressure swing（∆Pes） | At baseline and 15 minutes after each adjustment of the cisatracurium dose.
train train of four count (TOF-count) | At baseline and 15 minutes after each adjustment of the cisatracurium dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Affiliated to Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Force ADT, Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS: Acute respiratory distress syndrome: the Berlin Definition. JAMA 2012, 307(23):2526-2533. 2. Papazian L, Forel JM, Gacouin A, et al. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010;363(12):1107-1116. 3. Papazian L, Forel JM, Gacouin A, et al. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010;363(12):1107-1116. 4. Doorduin J, Nollet JL, Roesthuis LH, et al. Partial Neuromuscular Blockade during Partial Ventilatory Support in Sedated Patients with High Tidal Volumes. Am J Respir Crit Care Med. 2017;195(8):1033-1042. doi:10.1164/rccm.201605-1016OC 5. Guervilly C, Bisbal M, Forel JM et al (2017) Effects of neuromuscular blockers on transpulmonary pressures in moderate to severe acute respiratory distress syndrome. Intensive Care Med 43:408-418.17. Bouju P, Tadié JM, Barbarot N, et al. Clinical assessment and train-of-four measurements in critically ill patients treated with recommended doses of cisatracurium or atracurium for neuromuscular blockade: a prospective descriptive study. Ann Intensive Care. 2017;7(1):10. 6. Thompson Bastin ML, Smith RR, Bissell BD, et al. Comparison of fixed dose versus train-of-four titration of cisatracurium in acute respiratory distress syndrome. J Crit Care. 2021;65:86-90. 7. Hraiech S, Forel JM, Guervilly C, et al. How to reduce cisatracurium consumption in ARDS patients: the TOF-ARDS study. Ann Intensive Care. 2017;7(1):79.